CLINICAL TRIAL: NCT03739658
Title: Acute Effects of Cognitive Based Neuromuscular Education and Game Based Education on the Balance and Performance of Healthy Young Football Players
Brief Title: Acute Effects of Two Different Trainings on Balance and Performance in Young Footballers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murat EMİRZEOĞLU (Other)
Responsible Party: Sponsor-Investigator, Murat EMİRZEOĞLU, Research assistant, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-48
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Sports Physical Therapy
Keywords: Sports; Athletic Injuries; Exercise
MeSH Terms: conditions — Athletic Injuries; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Based Neuromuscular Education (Experimental): It will be applied for one hour. There are individual and partner parts. For example, in this training, the athlete will throw the tennis ball up and down on one foot.
  Interventions: Other: Education
- Game Based Education (Experimental): It will be applied for one hour. There are individual and partner parts. The active game will be played using the Xbox game console and the kinect sensor.
  Interventions: Other: Education
- Control Group (No Intervention): You will not receive any training. Athletes who continue their training as athletes in the other group.

INTERVENTIONS:
Other: Education — Cognitive-Based Neuromuscular Training has the content of focusing on different tasks at the same time and coordinating on neuromuscular functions as well as football-specific movements. Game-Based Training (OTE), which includes football, tennis, bowling, shooting, racing and climbing games, consists of active video games of game consoles, which are frequently used among young people.
  Arms: Cognitive Based Neuromuscular Education; Game Based Education

SUMMARY:
The aim of this study is to investigate the acute effect of two different training on the balance and performance of healthy young football players. Cognitive-Based Neuromuscular Education (CBNE) will be applied to one group and Game Based Education (GBE) will be applied to the other group. In addition to study groups, there will also be a control group. Individuals will be randomly placed in groups. Sociodemographic data will be recorded at the beginning for all athletes. Then the first measurements of dynamic balance and performance will be taken. Star Balance Excursion Test will be used to assess the dynamic balance. Measurements shall be taken in 8 directions including anterior (A), anterolateral (AL), lateral (L), posterolateral (PL), posterior (P), posteromedial (PM), medial (M) and anteromedial (AM) for the right and left sides. Performance will be evaluated by Speed Dribbling test. After the first measurements, two study groups will be trained. The control group will spend this time relaxing. After the trainings, the final measurements will be taken.

Purposes The primary purpose; The aim of this study was to investigate the acute effect of CBNE and GBE on dynamic balance and performance in healthy young football players.

Secondary objectives; The aim of this study is to investigate the relationship between dynamic balance and performance in healthy young football players.

hypotheses H0: In healthy young soccer players, CBNE and / or GBE has no acute effect on balance.

H0: In healthy young soccer players, CBNE and / or GBE has no acute effect on performance.

H1: CBNE and / or GBE have an acute effect on balance in healthy young football players.

H2: CBNE and / or GBE have an acute effect on performance in healthy young football players.

ELIGIBILITY:
Inclusion Criteria:

* To be playing active football for at least three years
* Males

Exclusion Criteria:

* Those with orthopedic, neurological or congenital problems
* Those who have experienced injuries that affect balance and performance in the last 6 months
* Individuals staying more than two weeks away from sport in the last three months

Ages: 15 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Balance | 45 minute
  Star Excursion Balance Test (cm)
Performance | 30 minute
  Speed Dribbling Test (sec)

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Ülger, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe Üniversitesi, Ankara, Türkiye, Turkey (Türkiye)

REFERENCES:
- [Derived] Emirzeoglu M, Ulger O. The Acute Effects of Cognitive-Based Neuromuscular Training and Game-Based Training on the Dynamic Balance and Speed Performance of Healthy Young Soccer Players: A Randomized Controlled Trial. Games Health J. 2021 Apr;10(2):121-129. doi: 10.1089/g4h.2020.0051. Epub 2020 Nov 9. PMID 33170049